CLINICAL TRIAL: NCT03391167
Title: Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Cholecystectomy Patients; Randomised, Controlled Prospective Study
Brief Title: Ultrasound Guided Bilateral Erector Spinae Plane Block in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., Assistant Professor of Anesthesiology, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MaltepeU
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Controlled randomised blinded preospective study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Peroperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Interventions: Other: Standard Pain Followup and Monitorization
- ESP Block (Experimental): In addition to routine analgesic protocol; before anaesthesia induction; bilateral ultrasound guided erector spinae plane block (ESP) (intervention) will be performed via USG guidance at Th9 level.Standard Pain Followup and Monitorization will be performed.
  Interventions: Procedure: Ultrasound guided erector spinae plane block; Other: Standard Pain Followup and Monitorization

INTERVENTIONS:
Procedure: Ultrasound guided erector spinae plane block — A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to T9 spinous process. The erector spinae muscles will be identified superficial to the tip of T9 transverse process. The patient's skin will be anesthetized with 2% lidocaine. A 17-gauge 8-cm needle will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of 0.375% bupivacaine will be injected (maximum of 3mg/kg).
  Arms: ESP Block
Other: Standard Pain Followup and Monitorization — Numeric Rating Scale (NRS) pain score will be recorded from 20th minute in recovery room followed by 1.-3.-6.-12.-18.-24.hours. Intravenous meperidine administration at 0.5 mg / kg rescue analgesia was determined in patients with a NSR score of 6 and over in the postoperative collection room. It is planned that the patient will continue to follow the hourly NRS score in ward. Intramuscular diclofenac will be administered in this period if NRS 6 and if it is over, intravenous 0.5 mg / kg meperidine will be administered if NRS score is 6 or more after 2 hours. Salvage analgesic needs and times will be noted in detail, and the use of rescue analgesics, as well as NRS scores at designated hours, will be kept in a statistical evaluation.

SUMMARY:
This study will define the postoperative analgesic effect of ESP block via amount of patient-controlled analgesia (PCA) and postoperative analgesic consumption (such as routinely and rescue analgesics) and compare the control group in patients having laparoscopic Cholecystectomy .

DETAILED DESCRIPTION:
Laparoscopic interventions are considered as minimally invasive procedures. They have both cosmetic and open surgery advantages in terms of surgical stress. Laparoscopic cholecystectomy is the most commonly performed laparoscopic upper abdominal procedure. After this procedure, patients often complain of excessive pain. Non-steroidal anti-inflammatory agents and opioids are used for postoperative analgesia. In addition, in the past decade, in the guideline of ultrasonography, peripheral block types with analgesic activity have been described in laparoscopic cholecystectomies as well as in many operations on the development of regional anesthesia and analgesia techniques. It was reported that transverse abdominis plane (TAP) block provided effective analgesia in these cases in the first ultrasonography guideline of petit triangle region in 2010. Later studies on TAP block activity, drug doses and concentrations in laparoscopic cholecystectomies have been conducted. There are also publications indicating that TAP block has been applied to the subcostal region for more effective analgesia. The ESP block is a new block for the treatment of thoracic neuropathic pain. In the following process; ESP block thoracic and breast surgery, bariatric surgery, and upper abdominal surgeons have also been reported to provide effective postoperative analgesia .

The standard practice for post-operative pain management for laparoscopic cholecystectomy in Maltepe University Hospital consists of routine intravenous analgesic and rescue analgesics and in combination with patient-controlled analgesia (PCA).

Given the importance of providing adequate analgesia in upper abdomen surgery and lack of consensus amongst surgeons and anesthesiologists for the optimal analgesic technique, the investigators are proposing a prospective observational study to examine the analgesic efficacy of the ESP block in laparoscopic cholecystectomy as a potential analgesic technique. The investigators are hoping the results of this study will provide framework for future larger comparative studies.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic Cholecystectomy, ASA status 1-2

Exclusion Criteria:

* Patient refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding diathesis
* Use of any anti-coagulants
* Inability to provide informed consent
* Severe kidney or liver disease
* Inability to operate PCA system
* Patient with psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, M.D., Study Director — Maltepe University Faculty of Medicine; Mahmut kapaklı, ass prof, Principal Investigator — maltepe universitesi
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016